CLINICAL TRIAL: NCT03985527
Title: Transvenous Nerve Stimulation Study (Janus Study)
Brief Title: Janus Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Respicardia, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CR1389
Record Dates: First submitted 2019-06-07; First posted 2019-06-13 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Sleep Apnea Syndromes
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Intervention Model Description: This is an acute, prospective, non-randomized, single arm IDE feasibility study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Transvenous nerve stimulation (Experimental)
  Interventions: Device: Transvenous nerve stimulation

INTERVENTIONS:
Device: Transvenous nerve stimulation — Acute transvenous nerve stimulation during a commercial implant of remedē® System or commercial transvenous cardiac device (de novo pacemaker or implantable cardiac defibrillator).

SUMMARY:
The purpose of this feasibility study is to assess whether an alternative transvenous lead location affects respiration and airway physiology during a commercial remedē® System or commercial transvenous cardiac device (de novo pacemaker or implantable cardiac defibrillator) implant procedure.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 years old
* Subject with moderate to severe central sleep apnea is undergoing a de novo commercial remedē® System implant procedure or other de novo transvenous cardiac implantable device procedure including a pacemaker or an implantable cardiac defibrillator
* Subject is willing and able to give informed consent

Exclusion Criteria:

* Subject is unable or unwilling to participate with study procedures or in the investigator's opinion is medically unstable for the procedure (Medically unstable is defined as when a patient is expected to have worsening health status if additional procedure time is needed)
* Subject is pregnant or planning to become pregnant (all women with childbearing potential must have a negative pregnancy test within 7 days prior to the implant)
* Subject is known to be allergic to radio opaque dye which cannot safely be pre-treated per the investigator
* Subject has body mass index (BMI) > 40 kg/m2 at the time of implant
* Subject has had prior neck surgery
* Previous or currently implanted upper airway stimulation device
* Subject has had prior oral cavity surgery that may interfere with breathing
* Subject has significant upper airway-related anatomic anomaly
* Subject is enrolled in concurrent study that may confound the results of this study
* Subject is taking muscle relaxant medication unless approved by the site implanter and ZOLL Respicardia clinical staff
* Subject has evidence of nerve weakness/paresis/paralysis or a neurologic disorder that involves the tongue

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2020-01-09 (Actual); Primary Completion 2025-12-12 (Actual); Study Completion 2025-12-12 (Actual)

PRIMARY OUTCOMES:
Changes in respiration and airway physiology | During procedure (immediately post-stimulation)
  The primary objective is to assess acute changes in respiration and airway physiology during the respiration cycle during a commercial remedē® System or commercial transvenous cardiac device (de novo pacemaker or implantable cardiac defibrillator) implant.

CONTACTS AND LOCATIONS:
Overall Officials: Kathy A McPherson, RN, MSN, Study Director — Respicardia, Inc.
Locations (3):
- United States (3):
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Bryn Mawr Medical Specialists Association, Bryn Mawr, Pennsylvania

IPD SHARING:
Plan to Share IPD: No